CLINICAL TRIAL: NCT04631445
Title: Randomized Phase II Trial of Two Different Nutritional Approaches for Patients Receiving Treatment for Their Advanced Pancreatic Cancer
Brief Title: Study Evaluating the Ketogenic Diet in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Drug Development (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TD2-PDAC-KETO-001
Record Dates: First submitted 2020-10-26; First posted 2020-11-17 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Metastatic Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Ketogenic Diet; Keto Diet
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Ketogenic diet with standard of care chemotherapy versus non-ketogenic diet with standard of care chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic (KD) + Triplet (Experimental): Ketogenic diet plus nab-paclitaxel 125 mg/m2, cisplatin 25 mg/m2, and gemcitabine 1000 mg/m2 all administered intravenously (IV) on Days 1 and 8 every 21 days.
  Interventions: Other: Ketogenic Diet
- Non-ketogenic + Triplet (No Intervention): Non-ketogenic diet plus nab-paclitaxel 125 mg/m2, cisplatin 25 mg/m2, and gemcitabine 1000 mg/m2 all administered intravenously (IV) on Days 1 and 8 every 21 days.

INTERVENTIONS:
Other: Ketogenic Diet — Ketogenic diet (KD) will consist of macros: dietary carbohydrates restricted to < 30 g/day; daily protein intake will be targeted to 1.5 g/kg/day (targeted to ideal body weight).
  Arms: Ketogenic (KD) + Triplet

SUMMARY:
This study will evaluate the effects of the ketogenic diet in patients with metastatic pancreatic cancer while receiving chemotherapy.

DETAILED DESCRIPTION:
A randomized, phase II trial designed to evaluate the progression free survival in patients with metastatic pancreatic cancer on triplet therapy (nab-paclitaxel + gemcitabine + cisplatin) while on ketogenic diet or non-ketogenic diet. This study also aims to compare the changes in serum metabolites and quality of life between the two arms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age; male or female.
2. Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma, not previously treated for their metastatic disease.
3. Capable of providing informed consent and complying with trial procedures.
4. Karnofsky Performance Status (KPS) of ≥ 70%.
5. Life expectancy ≥ 12 weeks.
6. Measurable tumor lesions according to RECIST 1.1 criteria.
7. <Grade 2 pre-existing peripheral neuropathy per NCI CTCAE, Version 5.0.
8. Patient has acceptable coagulation status as indicated by an INR ≤1.5 times institutional upper limit of normal (ULN). Patients on anticoagulation can be included at the discretion of the investigator.
9. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count ≥1,500/mm3
   * Platelet concentration ≥100,000/mm3 with no platelet transfusions within 7 days prior to laboratory sample
   * Hemoglobin ≥ 9.0g/dL (PRBCs may be given to meet this criteria)
   * Hematocrit level ≥ 27%
   * Total bilirubin within 1.25 x ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 times upper limit of normal (if liver metastases are present, then ≤ 5 x ULN is allowed)
   * Serum creatinine < 1.5 mg/dL.
10. Patient must have a Smartphone or computer in order to work with Virta
11. Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

    1. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting IP therapy (including dose interruptions), and while on study medication or for a longer period if required by local regulations following the last dose of IP; and
    2. Have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
12. Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following discontinuation from study treatment, even if he has undergone a successful vasectomy.

    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

Exclusion Criteria:

1. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of their metastatic pancreatic disease. Prior treatment in the adjuvant setting with chemotherapy and radiation are allowed, provided at least 6 months have elapsed since completion of the last therapy and recurrence and no lingering toxicities are present (this will be first line treatment for metastatic disease).
2. Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
3. History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for ≥ 2 years.
4. Uncontrolled intercurrent illness, including but not limited to New York Heart Association Class III or IV, myocardial infarction within the past 6 months, or unstable arrhythmia.
5. Known infection with HIV, hepatitis B, or hepatitis C.
6. Active, uncontrolled bacterial, viral, or fungal infections, requiring systematic therapy.
7. Major surgery within 4 weeks prior to study entry. (Port-a-cath may be inserted during this time period).
8. Any condition in the opinion of the principal investigator that might interfere with the patient's participation in the study or in the evaluation of the study results.
9. Any condition in the opinion of the principal investigator that is unstable and could jeopardize the patient's participation in the study.
10. Unwillingness or inability to comply with procedures required in this protocol, including unwillingness to follow a ketogenic diet.
11. Severe malnutrition or body mass index (BMI) < 18.
12. Albumin < 3.0 g/dL.
13. History of Type 1 diabetes.
14. History of diabetic ketoacidosis (DKA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival per RECIST 1.1 | 36 months
  Progression-free survival (PFS) is defined as the time from randomization to first documentation of objective tumor progression or to death due to any cause.

SECONDARY OUTCOMES:
To compare the number of responses by RECIST 1.1 | 36 months
  To compare the number of complete responses/partial responses as defined by CT scan using the Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) and CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9) down to normal limits (from at least > 2X ULN).
To compare the disease control rate using the Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1). | 36 months
  (Partial Response + Complete Response + Stable Disease for at least 9 weeks)
Cancer Biomarkers | 36 months
  Change in CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9)
Cancer Biomarkers returning to normal | 36 months
  Rates of normalization of CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9)
Change in BMI | 36 months
  To compare the average weight (kg), using BMI calculation (BMI = weight (kg) / height (m2))
Compare insulin levels | 36 months
  To compare average insulin levels
To compare the average HbgA1c level | 36 months
  To compare the average HbgA1c levels
To compare changes in serum metabolites | 36 months
  To compare changes in serum metabolites
To compare quality of life between arms via the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire QLC-C30 (EORTC QLQ-C30) assessment. | 36 months
  Higher scores in the quality of life on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire QLC-C30 (EORTC QLQ-C30) assessment may show a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Norton, MBA PhD, Study Director — Translational Drug Development
Locations (6):
- United States (6):
  - Honor Health, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Nuvance Health-Danbury Hospital, Danbury, Connecticut
  - Nuvance Health, Norwalk, Connecticut
  - Tennessee Oncology, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang L, TeSlaa T, Ng S, Nofal M, Wang L, Lan T, Zeng X, Cowan A, McBride M, Lu W, Davidson S, Liang G, Oh TG, Downes M, Evans R, Von Hoff D, Guo JY, Han H, Rabinowitz JD. Ketogenic diet and chemotherapy combine to disrupt pancreatic cancer metabolism and growth. Med. 2022 Feb 11;3(2):119-136. doi: 10.1016/j.medj.2021.12.008. PMID 35425930